CLINICAL TRIAL: NCT05648539
Title: Effect of Music Therapy in Mental Subhealth: A Randomized Controlled Trial
Brief Title: Effect of Music Therapy in Mental Subhealth (EMTMS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81725005-4
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Depression, Anxiety
Keywords: Music Therapy; Depression, Anxiety; Acoustic features
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The clinical response of the music therapy (Experimental): To assessthe efficacy of music therapy of MT group compared to Waiting group in mental subhealth.
  Interventions: Device: The mini apps named "SOUL GYM" on the Wechat
- The alterations of acoustic features in the music therapy (Experimental): To understand the possible biological mechanism underlying the efficacy of music therapy by analyzing alterations of acoustic features.
  Interventions: Device: The mini apps named "SOUL GYM" on the Wechat

INTERVENTIONS:
Device: The mini apps named "SOUL GYM" on the Wechat — Music Therapy can make peoples gradually relax via relaxing and soothing music, and regulate individual psychological emotions through the influence of music on individuals' cerebral cortex, hypothalamus and limbic system, further improve the mood of daily tension and anxiety.

SUMMARY:
Mental health is increasingly at the forefront of concerns, especially since the start of COVID-19 pandemic. However, not all individuals under mental subhealth need pharmaceutical treatment. Music Therapy (MT) can make peoples gradually relax via relaxing and soothing music, and regulate individual psychological emotions through the influence of music on individuals' cerebral cortex, hypothalamus and limbic system, further improve the mood of daily tension and anxiety.

This study adopted randomized clinical trials design, with two groups of MT group and Waiting group both under mental subhealth. The MT group received music therapy and routine activities, while the Waiting group received music therapy after the therapy of MT group. Data collections were performed by trained, certified, and qualified personnel. The study aims to provide that MT is an effective intervention way to alleviate the mental subhealth state in the future.

DETAILED DESCRIPTION:
This study is a double-blind randomized controlled trial aiming at assessing the efficacy of MT compared to Waiting group in mental subhealth. Participants will be assigned randomly (1:1) to MT group and Waiting group. All the participants will be treated with 12 sessions (3 sessions per week), 30 minutes each time, and conducted for 4 weeks. The MT group received music therapy between 1st-4th week, and the Waiting group received music therapy between 5th-8th week. Pre-MT (baseline) and post-MT (4th week), two group performed symptom assessment and voice data collection (poetry readings). The MT is mainly divided into three stages, and each stage has a topic. The topic of each stage as follow: ① physical and mental relaxation stage: learning the whole body and mind relaxation mode from breathing to muscle; ② nature imagination stage: guiding music imagination; ③ internal self-exploration: excavating the positive experience and positive potential of the listener and adopting resource orientation for psychological intervention. The purposes of the present study are to: 1) evaluate the clinical response the MT in mental subhealth. 2) further understand the possible biological mechanism underlying the efficacy of MT by analyzing alterations of acoustic features.

ELIGIBILITY:
Inclusion Criteria:

A total of > 5 on PHQ-9 or a total of > 5 on GAD-7

Exclusion Criteria:

Acute suicidal thoughts, With a severe or potentially confounding psychiatric disorder (e.g. psychosis, substance misuse).

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-19 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms assessed by the Patient Health Questionnaire-9 (PHQ-9; range: 0-27) at week 4. | Baseline and week 4.
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-27) depression.
Change from baseline in anxiety symptoms assessed by the Generalized Anxiety Disorder-7 (GAD-7, range: 0-21) at week 4. | Baseline and week 4.
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Change from baseline in insomnia symptoms assessed by the Insomnia Severity Index (ISI; range: 0-28) at week 4. | Baseline and week 4.
  The total scores of these questionnaires were interpreted as follows: normal (0-7), mild (8-14), moderate (15-21), and severe (22-28) insomnia.
Change from baseline in perceived stress assessed by the Perceived Stress Scale-14 (PSS-14; range: 0-56) at week 4. | Baseline and week 4.
  The total scores of these questionnaires were interpreted as follows: normal (0-28), moderate (29-42), severe (43-56).

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Study Chair — Affiliated Nanjing Brain Hospital, Nanjing Medical University
Locations (1):
- Affiliated Nanjing Brain Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang L, Zhu Y, Zheng Z, Ma H, Cai X, Yang H, Wang F. Music Therapy Modulates Abnormal Brain Networks and Alleviates Anxiety Symptoms in University Students: An fNIRS Study. Depress Anxiety. 2025 Nov 20;2025:7906429. doi: 10.1155/da/7906429. eCollection 2025. PMID 41321481